CLINICAL TRIAL: NCT04254081
Title: Addition of Buprenorphine to Paracervical Block Prior to Osmotic Dilator Insertion for Dilation and Evacuation: A Randomized Controlled Trial
Brief Title: Addition of Buprenorphine to Paracervical Block for Pain Control During Osmotic Dilator Insertion
Acronym: ABCD&E
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Sheila Mody, Associate Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 192033
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Procedural Pain; Buprenorphine; Adjuvants, Anesthesia; Dilation and Evacuation; Analgesics
Keywords: Abortion; Osmotic dilators; Cervical preparation
MeSH Terms: conditions — Pain, Procedural; Dilatation, Pathologic | interventions — Buprenorphine; Lidocaine

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo controlled trial with stratified block randomization based on vaginal parity (vaginally nulliparous versus vaginally multiparous). Vaginal parity may influence pain during osmotic dilator insertion and thus the participants will be evenly distributed between strata.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A clinician who will not be administering the paracervical block will open the designated sealed sequentially numbered opaque randomization envelope containing computer generated randomization code and prepare the designated paracervical block into two 10 mL syringes. The syringes used to prepare the medication will be identical between study groups and the solutions will appear visually identical. A different clinician blinded to the treatment group will perform the standardized procedure for osmotic dilator insertion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine 0.15mg + 1% lidocaine paracervical block (Experimental): Paracervical block with 18mL of 1% lidocaine buffered with 2 mL 8.4% sodium bicarbonate plus 0.15mg of buprenorphine
  Interventions: Drug: Buprenorphine 0.15 MG
- 1% lidocaine paracervical block (Placebo Comparator): Paracervical block with 18 mL of 1% lidocaine buffered with 2 mL 8.4% sodium bicarbonate
  Interventions: Drug: Lidocaine 1% Injectable Solution

INTERVENTIONS:
Drug: Buprenorphine 0.15 MG — Buprenorphine 0.15mg solution will be added to a 20mL 1% buffered lidocaine solution (paracervical block) which will be administered in the paracervical space prior to osmotic dilator insertion.
  Arms: Buprenorphine 0.15mg + 1% lidocaine paracervical block
Drug: Lidocaine 1% Injectable Solution — 20mL of 1% buffered lidocaine solution (paracervical block) will be administered in the paracervical space prior to osmotic dilator insertion.
  Arms: 1% lidocaine paracervical block

SUMMARY:
Cervical preparation with osmotic dilators is commonly used prior to dilation and evacuation (D&E) procedures to decrease the risk of complications. Women have described the pain of osmotic dilator insertion as moderate to severe yet there have been few studies aimed at addressing pain during and after osmotic dilator insertion. In addition to the discomfort during insertion, pain after osmotic dilator insertion peaks at 2 hours post-insertion with use of a lidocaine paracervical block. One randomized trial found that use of a paracervical block with 1% buffered lidocaine decreased pain with osmotic dilator insertion compared to a sham block. There are adjunct treatments to optimize analgesia with local anesthetics at a variety of anatomic locations. Buprenorphine, a partial mu-opioid receptor agonist, has been found to increase the quality of the anesthetic at the time of administration and increase the duration of nerve block analgesia at several anatomic sites, though has never been studied as an adjunct in a paracervical block. This has been used extensively in orthopedic surgery with significant prolongation of the local anesthetic effect by almost threefold in some studies.

Primary Aim: To compare the mean pain score at the time of osmotic dilator insertion among women randomized to a 1% lidocaine and buprenorphine paracervical block compared to a 1% lidocaine paracervical block alone.

Secondary Aim: To compare the mean pain score 2 hours after osmotic dilator insertion among women randomized to a lidocaine and buprenorphine paracervical block compared to a lidocaine paracervical block alone.

The investigators hypothesize that in patients undergoing osmotic dilator insertion in preparation for dilation and evacuation, the addition of buprenorphine 0.15mg to a 1% lidocaine paracervical block will be associated with lower mean pain scores at time of osmotic dilator insertion compared to women who receive a 1% lidocaine paracervical block alone.

DETAILED DESCRIPTION:
Dilation and evacuation (D&E) is the most common method of second trimester abortion in the United States. Cervical preparation prior to the procedure is essential in order to allow passage of operative instruments and pregnancy tissue safely through the cervix and to decrease the risk of complications. In the second trimester, cervical preparation is typically achieved with placement of osmotic dilators prior to the procedure. Women have described the pain of osmotic dilator insertion as moderate to severe yet there have been few studies aimed at addressing pain during osmotic dilator insertion. A lidocaine paracervical block is commonly used for pain control during other gynecologic procedures including procedures involving cervical dilation like dilation and curettage. One randomized controlled trial found that use of a paracervical block with 1% lidocaine decreased pain with osmotic dilator insertion compared to a sham block. Because the dilators slowly expand after insertion, there is continued discomfort for several hours after placement. Research has shown that pain after osmotic dilator insertion peaks at 2 hours post-insertion with use of a lidocaine paracervical block and a local anesthetic is not sufficient to provide lasting pain relief. Systemic medications, such as gabapentin and narcotic analgesics have been studied to treat post-insertional dilator pain, however these treatments have not been shown to be effective.

There are many adjunct treatments to optimize the duration of local analgesia from a peripheral nerve block. Buprenorphine, a partial mu-opioid receptor agonist, is a high potency, lipophilic opioid and has a high binding capacity for the mu-opioid receptor. Because of the high binding capacity, buprenorphine has the longest duration of action of all opioids. When administered perineurally in combination with a local anesthetic, buprenorphine has been found to drastically increase the duration of analgesia at several anatomic sites, including axillary and subclavian brachial plexus blocks and infragluteal sciatic nerve blocks. With the addition of buprenorphine at doses of 0.15 - 0.3mg, there is significant prolongation of the anesthetic sensory blockade up to three times the duration of the local anesthetic alone. The use of perineural buprenorphine is well established for postoperative analgesia. Buprenorphine itself also has local anesthetic properties. Buprenorphine blocks voltage gated sodium channels and inhibits C-fiber action potentials, thereby contributing to an analgesic effect. Buprenorphine not only prolongs the duration of local anesthetic effect but also improves the analgesic properties when administered in a perineural block.

The addition of buprenorphine to a perineural local anesthetic has not been studied in a paracervical block. This study will be the first trial to assess the efficacy of buprenorphine to provide analgesia for a gynecologic procedure. This medication has the additional benefit of providing long lasting pain relief for procedures that cause continued discomfort after the end of the procedure. The investigators hypothesize that the addition of 0.15mg of buprenorphine to a lidocaine paracervical block will improve pain during osmotic dilator insertion and provide continued pain relief several hours after osmotic dilator insertion. If this intervention proves to provide better pain control than a lidocaine paracervical block alone, it would be an intervention for women during a painful clinic procedure.

A total of 114 women undergoing D&E who require cervical preparation with osmotic dilators will be randomized to one of two study groups: (1) paracervical block with 20mL of 1% buffered lidocaine or (2) paracervical block with 20mL of 1% buffered lidocaine plus 0.15mg of buprenorphine. Participants, clinicians performing the procedure, and study personnel administering questionnaires will be blinded to study assignment. Participants will rate their level of pain on an 11-point numeric rating scale (NRS) during the insertion of osmotic dilators and at several time points after insertion. The primary outcome is to compare the median pain score at the time of osmotic dilator insertion in women randomized to a 1% lidocaine and buprenorphine paracervical block compared to a 1% lidocaine paracervical block alone. Secondary outcomes are to compare the median pain score 2 hours after osmotic dilator insertion; to assess overall narcotic and ibuprofen use after osmotic dilator placement and before dilation and evacuation procedure; to assess opioid related side effects; and to determine patient satisfaction with pain control during and after osmotic dilator insertion.

Primary Hypothesis: The addition of buprenorphine 0.15mg to a paracervical block using 1% lidocaine will be associated with a lower median pain score on the NRS at time of osmotic dilator insertion compared to women who receive a lidocaine paracervical block alone.

Secondary Hypothesis: The addition of buprenorphine 0.15mg to a paracervical block using 1% lidocaine will be associated with a lower median pain score on the NRS 2 hours after osmotic dilator insertion compared to women who receive a lidocaine paracervical block alone.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 14 0/7 weeks to 23 6/7 weeks at time of osmotic dilator insertion
* Require cervical preparation with placement of osmotic dilators
* At least 18 years of age
* Fluent in English or Spanish

Exclusion Criteria:

* Same day dilation and evacuation procedure
* Request for sedation during osmotic dilator insertion
* Liver disease
* Allergy to buprenorphine, lidocaine, or ibuprofen
* Narcotic or opioid medication use in the preceding 24 hours
* Use of recreational/illicit medications in the preceding 24 hours
* Currently incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Economou, MD, Principal Investigator — UC San Diego Health; Sheila K Mody, MD, MPH, Principal Investigator — UC San Diego Health
Locations (1):
- University of California San Diego Health, San Diego, California, United States

REFERENCES:
- [Background] Schivone GB, Lerma K, Montgomery C, Wright P, Conti JA, Blumenthal PD, Shaw KA. Self-administered lidocaine gel for local anesthesia prior to osmotic dilator placement: a randomized trial. Contraception. 2019 Mar;99(3):148-151. doi: 10.1016/j.contraception.2018.11.013. Epub 2018 Nov 27. PMID 30500336
- [Background] Soon R, Tschann M, Salcedo J, Stevens K, Ahn HJ, Kaneshiro B. Paracervical Block for Laminaria Insertion Before Second-Trimester Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2017 Aug;130(2):387-392. doi: 10.1097/AOG.0000000000002149. PMID 28697113
- [Background] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724
- [Background] Creinin MD, Schimmoeller NR, Matulich MC, Hou MY, Melo J, Chen MJ. Gabapentin for pain management after osmotic dilator insertion and prior to dilation and evacuation: A randomized controlled trial. Contraception. 2020 Mar;101(3):167-173. doi: 10.1016/j.contraception.2019.12.001. Epub 2020 Jan 10. PMID 31927028
- [Background] Kosel J, Bobik P, Tomczyk M. Buprenorphine--the unique opioid adjuvant in regional anesthesia. Expert Rev Clin Pharmacol. 2016;9(3):375-83. doi: 10.1586/17512433.2016.1141047. Epub 2016 Jan 28. PMID 26758991
- [Background] Bailard NS, Ortiz J, Flores RA. Additives to local anesthetics for peripheral nerve blocks: Evidence, limitations, and recommendations. Am J Health Syst Pharm. 2014 Mar 1;71(5):373-85. doi: 10.2146/ajhp130336. PMID 24534592
- [Background] Swain A, Nag DS, Sahu S, Samaddar DP. Adjuvants to local anesthetics: Current understanding and future trends. World J Clin Cases. 2017 Aug 16;5(8):307-323. doi: 10.12998/wjcc.v5.i8.307. PMID 28868303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multi-site, randomized, double-blind controlled trial conducted from May 2020-May 2021. Participants presenting for dilation and evacuation who required osmotic dilators for cervical preparation were randomized 1:1 to receive a 1% buffered lidocaine PCB or a 1% buffered lidocaine + 0.15mg buprenorphine PCB.
Period: Overall Study
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block
Started | 28 | 29
Completed | 28 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 4 | 6 | 10
  Race/Ethnicity: Black or African American | 1 | 1 | 2
  Race/Ethnicity: Hispanic or Latina | 19 | 15 | 34
  Race/Ethnicity: Asian | 1 | 5 | 6
  Race/Ethnicity: Other or multiracial | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at the Time of Osmotic Dilator Insertion
Description: Median pain score on a 0 (no pain) to 10 (worst pain) numeric rating scale at the time of osmotic dilator insertion
Time Frame: Assessed immediately after last dilator inserted
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block
Number analyzed (Participants) | 28 | 29
score on a scale | 3.5 [1 to 6] | 4.0 [2 to 7]

2. Secondary Outcome: Pain Score 2 Hours After Osmotic Dilator Insertion
Description: Median pain score on a 0 (no pain) to 10 (worst pain) numeric rating scale 2 hours after osmotic dilator insertion assessed via text message
Time Frame: 2 hours after osmotic dilator insertion
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block
Number analyzed (Participants) | 28 | 29
score on a scale | 3 [1 to 5] | 3.5 [1 to 5]

3. Secondary Outcome: Pain Score 1 Hour After Osmotic Dilator Insertion
Description: Median pain score on a 0 (no pain) to 10 (worst pain) numeric rating scale 1 hour after osmotic dilator insertion assessed via text message
Time Frame: 1 hour after osmotic dilator insertion
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block
Number analyzed (Participants) | 28 | 29
score on a scale | 2 [1 to 3] | 3.5 [1.75 to 5.25]

4. Secondary Outcome: Pain Score 6 Hours After Osmotic Dilator Insertion
Description: Median pain score on a 0 (no pain) to 10 (worst pain) numeric rating scale 6 hours after osmotic dilator insertion assessed via text message
Time Frame: 6 hours after osmotic dilator insertion
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block
Number analyzed (Participants) | 28 | 29
score on a scale | 3 [1.75 to 5.25] | 3 [0.5 to 4.5]

5. Secondary Outcome: Overall Satisfaction Scores
Description: To determine patient satisfaction with pain control during and after osmotic dilator insertion. This was assessed on the morning of D&E procedure. Participants following question and rated responses on a Likert scale:
  What was your overall satisfaction with the amount of pain control that you had during the procedure?
Time Frame: Morning of D&E procedure: after check-in, before D&E
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block
Number analyzed (Participants) | 28 | 29
Participants
  Very Satisfied | 14 | 13
  Satisfied | 9 | 14
  Slightly Satisfied | 3 | 0
  Slightly dissatisfied | 2 | 1
  Dissatisfied | 0 | 0
  Very dissatisfied | 0 | 1

ADVERSE EVENTS:
Time Frame: Day of procedure from time of enrollment to time of discharge, approximately 36 hours.
Arm/Group | Buprenorphine 0.15mg + 1% Lidocaine Paracervical Block | 1% Lidocaine Paracervical Block
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04254081/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04254081/ICF_001.pdf